CLINICAL TRIAL: NCT01490021
Title: Influence of Repetitive Transcranial Magnetic Stimulation (rTMS) Challenge on Cognitive and Functional Magnetic Resonance Imaging Markers in Healthy Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped for scientific reasons. Another study with a new design is in course of authorization and implementation
Sponsor: Qualissima (Other)
Collaborators: Pharmacog's project (IMI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: WP1P002
Record Dates: First submitted 2011-11-28; First posted 2011-12-12 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: Healthy young men

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS/Active TBS (Experimental): A continuous Theta-Burst Stimulation (TBS) protocol will be applied over the left dorsolateral prefrontal cortex. Three stimuli at 50Hz, 80% of individual Motor Threshold will be repeated every 200ms for 40sec (Galea et al., 2010; Oberman and Pascual-Leone, 2009).
  Interventions: Procedure: rTMS/Active TBS
- rTMS/Placebo TBS (Placebo Comparator): rTMS/Placebo TBS
  Interventions: Procedure: rTMS/Placebo TBS

INTERVENTIONS:
Procedure: rTMS/Active TBS — A continuous Theta-Burst Stimulation (TBS) protocol will be applied over the left dorsolateral prefrontal cortex. Three stimuli at 50Hz, 80% of individual Motor Threshold will be repeated every 200ms for 40sec (Galea et al., 2010; Oberman and Pascual-Leone, 2009).
  Arms: rTMS/Active TBS
Procedure: rTMS/Placebo TBS — rTMS/Placebo TBS
  Arms: rTMS/Placebo TBS

SUMMARY:
Episodic and working memory processes are the most affected cognitive domains in Alzheimer's Disease (AD) and its early stage, Mild Cognitive Impairment (MCI). Transcranial Magnetic Stimulation (TMS) is a unique tool to interfere with cognitive processes by inducing "virtual and transient lesions", mimicking those observed in MCI. It has proven repeatedly its capacity to interfere with encoding-retrieval memory task. However, to date, only few imaging data exist on the cerebral pathways involved in encoding memory task. Moreover, the stability of TMS effects over time remains to be investigated. If proven to be a stable interfering challenge, TMS could be used to investigate the potential restoring effect of new medication in AD.

The study is the pilot study of a larger clinical trial which aims to prove the utility of rTMS as a potential model for prediction of clinical efficacy using a combination of cognitive and neuroimaging endpoints.

DETAILED DESCRIPTION:
Episodic and working memory processes are the most affected cognitive domains in Alzheimer's Disease (AD) and its early stage, Mild Cognitive Impairment (MCI). Transcranial Magnetic Stimulation (TMS) is a unique tool to interfere with cognitive processes by inducing "virtual and transient lesions", mimicking those observed in MCI. It has proven repeatedly its capacity to interfere with encoding-retrieval memory task. However, to date, only few imaging data exist on the cerebral pathways involved in encoding memory task. Moreover, the stability of TMS effects over time remains to be investigated. If proven to be a stable interfering challenge, TMS could be used to investigate the potential restoring effect of new medication in AD.

The study is the pilot study of a larger clinical trial which aims to prove the utility of rTMS as a potential model for prediction of clinical efficacy using a combination of cognitive and neuroimaging endpoints.

This pilot study specifically aims:

* to determine the cerebral region to stimulate using functional neuronavigation,
* to evaluate the effects of rTMS on behavioral and functional imaging data (functional Magnetic Resonance Imaging, fMRI)
* to investigate the stability of the TMS interfering effects by replicating the experimental day up to 4 times.

The study is composed of two parts:

* Part A: on Day 1, the subjects will perform the episodic memory task in the MRI scanner to determine individual main activations. The mean activation peak obtained by a group analysis will be used as the target coordinates during the part B. Two weeks later, on Day 2, the subjects will repeat the episodic memory task in the MRI scanner. The BOLD signal changes will be compared between Day 1 and Day 2 to investigate the stability of the activations elicited by the memory task.
* Part B: subjects will randomly be assigned to Group 1 or 2.

  * GROUP 1: The subjects will come on 4 different days. On each day, the subjects will perform the episodic memory task while being actively stimulated using rTMS over L-DLPFC and Vertex (control region) in random order and will undergo an fMRI session on Day 1 and Day 2. Later, they will undergo another set of behavioral tasks from the CANTAB battery and will be stimulated by rTMS using a placebo coil.
  * GROUP 2: The subjects will come on 4 different days. On each day, the subjects will perform the episodic memory task while being actively stimulated using rTMS over L-DLPFC and Vertex (control region) in random order and will undergo an fMRI session on Day 1 and Day 2. Later, they will undergo another set of behavioral tasks from the CANTAB battery and will be stimulated by rTMS using an active coil.

Total expected number of subjects:

34 subjects for the Parts A and B PART A: 10 subjects PART B: 24 subjects (12 per group)

ELIGIBILITY:
Inclusion Criteria:

Demography

1. Healthy male subjects aged between 18 and 40 years-old inclusive.
2. BMI between 18 kg/m2 to 29 kg/m2.
3. Education level: at least secondary.
4. Right-handed (Edinburgh Handedness Inventory).

   * Health status
5. The subjects is in good health on the basis of the medical interview (medical history, symptoms) and the physical examination, vital signs.
6. No history of psychiatric or neurological disorders as assessed by Structured Clinical Interview for DSM IV Disorders (SCID).
7. No history of concussion with loss of consciousness more than 20 min.
8. No history of drug or alcohol abuse.

   * Specific to the study
9. The subject can complete the neuropsychological test battery during the training session.

   * Regulations
10. The subject is able to read and understand the Information Form and comply with the protocol instructions and restrictions
11. The subject is covered by a social insurance
12. The subject have provided written informed consent

Exclusion Criteria:

* Medical history and clinical status

  1. History or presence of psychiatric illness (Psychiatric interview).
  2. History or presence of neurologic illness.
* General conditions 3. The subject, in the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any other reason.

  4. The subject participates in another clinical trial or is still being within a washout period of 1 month since last taking of a previous clinical trial, or subjects who have received more than 4500 Euros in the previous 12 months for participating in clinical trials.
* Specific to the study 5. Presence of metallic objects within the head. 6. Subjects with pacemaker. 7. Claustrophobia. 8. Individual and familial history of seizure. 9. Any medication listed in the safety guidelines published by the Safety of TMS Consensus Group (Rossi et al., 2009) will be forbidden.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Part A: Location of cerebral activities | Day 1
  Primary endpoints:
  The location of cerebral activities elicited by the retrieval session of the episodic memory task during fMRI will be the primary endpoint of PART A.
  PART A will assess task-elicited BOLD signal modifications and determine the target location coordinates and verify the stability of the BOLD signal responses over time and the stability of the target location
Part B: Outputs of the memory task | Change between Day 2 and Day 1
  Outputs: the number of correct answers during the retrieval blocks (Hit rates)and the number of false recognition of novel pictures (False Alarms rate).

SECONDARY OUTCOMES:
Part A: The outputs of the memory task | Day 1 and Day 2
  Memory task. The output of the task will be the number of correct answers during the retrieval blocks (i.e. correctly recognized images presented during the encoding blocks, Hits rate) and the number of false recognition of novel pictures (False Alarms rate).
Part B: Imaging and CANTAB tasks | Day 1, 2, 3 and 4
  Imaging (functional MRI): Modifications will be highlighted by changes in the Blood-Oxygen-Level Dependence (BOLD) signal patterns.
  CANTAB tasks:
  * CANTAB / Rapid Visual Information Processing (RVP) with outcome measures: latency, probabilities and sensitivity and hits, misses, false alarms and rejections;
  * CANTAB / Spatial Working Memory (SWM) with outcome measures: errors, strategy and latency measures.
  * CANTAB / Paired Associates Learning (PAL) with outcome measures: errors, number of trials required to locate the pattern(s) correctly, memory scores.

CONTACTS AND LOCATIONS:
Overall Officials: David Bartrés-Faz, Principal Investigator — Institut d'Investigacions Biomèdiques August Pi i Sunyer
Locations (1):
- IDIBAPS, Barcelona, Spain